CLINICAL TRIAL: NCT00982956
Title: Application of Computer-assisted Navigation in Total Knee Arthroplasty: A Randomized Pair-matched Double-blind Trial
Status: Completed | Type: Observational
Sponsor: Chinese PLA General Hospital (Other)
Other Study IDs: 2007023
Record Dates: First submitted 2009-09-22; First posted 2009-09-23 (Estimated); Last update posted 2009-09-23 (Estimated); Status verified 2009-09

CONDITIONS: Knee Arthritis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective

SUMMARY:
Objective:

The purpose of this study is to evaluate the application of computer-assisted navigation in Total Knee Arthroplasty (TKA ) by comparing it with conventional TKA.

Methods:

Gemini MK II implants (Link, Germany) were used. VectorVisionâ CT-free navigation system (BrainLab, Germany) was employed for the TKA. For each subject, computer-navigation TKA and the conventional TKA were separately performed on two knee joints. The operative method and order of the operations were decided on a randomized basis. All the patients and doctors conducting follow-up study and performing imaging measurement were blind to selection of the operation. Student t test was used for statistical analysis.

hypothesis: computer-assisted navigation system can significantly improve the accuracy of tibial and femoral cuts on coronal and sagittal planes.

ELIGIBILITY:
Inclusion Criteria:

* plan for simultaneous bilateral TKA.

Exclusion Criteria:

* plan for unilateral TKA.

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: the subjects who had been scheduled for simultaneous bilateral TKA,
Sampling Method: Probability Sample